CLINICAL TRIAL: NCT03996577
Title: Efficacy of Intravenous Infusion of Lidocaine in Sedation for ERCP: a Randomised Placebo-controlled Study
Brief Title: Intravenous Infusion of Lidocaine in ERCP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2019SDU-QILU-071
Record Dates: First submitted 2019-06-18; First posted 2019-06-25 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Sedation
Keywords: lidocaine propofol ercp
MeSH Terms: interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to controll group or lidocaine group. Participants of control group are given placebo while participants of lidocaine group are given lidocaine.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): the control group will be given the same volume of saline as the experimental group
  Interventions: Drug: placebo
- Experimental: lidocaine group (Experimental): the experimental group will be given l-1.5mg lidocaine and then 2mg/kg/h
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — the experimental group will be given 1-1.5mg/kg lidocaine and then 2mg/kg/h
  Other Names: Compound Lidocaine Hydrochloride Injiection
  Arms: Experimental: lidocaine group
Drug: placebo — the control group will be given the same volume of saline.
  Other Names: saline
  Arms: control group

SUMMARY:
Intravenous infusion of lidocaine significantly reduces propofol dose for ERCP and improve patients' recovery after ERCP.

DETAILED DESCRIPTION:
This study divide patients into two groups, one will be given lidocaine; another group was given placebo . to observe two groups of patients blood pressure, body movement, and propofol dosage , and the difference in operator satisfaction, and how many people need to give fentanyl again; and two groups of patients after the operation of the reaction, if there are dizziness, nausea, and other adverse reactions; finally, the differences of these two schemes in different populations were analyzed, and the rationalization and individualized medication will be put forward.

ELIGIBILITY:
Inclusion Criteria:Inpatients aged >18 years who were scheduled for ERCP at Qilu hospital.

Exclusion Criteria:

* Patients with ASA class 4 or 5,
* Patients with pre-existing hypoxaemia (SpO2<90%),
* Patients with hypotension (SBP<90mmHg)
* Patients with bradycardia (HR<50 bpm)
* patients with severe chronic renal failure (creatinine clearance<30 ml/min)
* patients with uncontrolled hypertension (systolic blood pressure>170 mm Hg, diastolic blood pressure>100 mm Hg)
* patients with pregnancy or lactation
* Patients hemodynamically unstable
* Patients unable to give informed consent
* Patients with a history of drug allergies;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-10-15 (Estimated); Study Completion 2019-11-15 (Estimated)

PRIMARY OUTCOMES:
propofol consumption difference between the two groups | half a year
  the total propofol dosage consumption between the two groups

SECONDARY OUTCOMES:
Safety assessed by the rate of hypoxia during the procedure Safety assessed by the rate of hypoxia during the procedure | half a year
  Hypoxia, defined as peripheral oxygen saturation <90% for >30 seconds
Safety assessed by the rate of hypotention during the procedure | half a year
  Hypotension, defined as systolic blood pressure <90 mmHg
Safety assessed by the rate of breadycardia during the procedure | half a year
  Bradycardia, defined as heart rate <50 beats/min
Safety assessed by the rate of required airway management during the procedure | half a year
  Required airway management such as jaw lifting, mask ventilation, or tracheal intubation in severe hypoxia Required airway management such as jaw lifting, mask ventilation, or tracheal intubation in severe hypoxia
Safety assessed by the rate of involuntary movement during the procedure | half a year
  Involuntary movements, defined as unconscious movements requiring restraint or severe limb movement interrupting the endoscopy procedure
endoscopists satisfaction assessed by the performer | half a year
  the endoscopists satisfacition score were assessed on a 0-10VAS after the procedure
patient satisfaction assessed by the patient | half a year
  the patient satisfacition score were assessed on a 0-10VAS 30mins after the procedure
pain socre after the ERCP | half a year
  pain were measured on a 0-10VAS at arrival in the recovery room ,30min later
fatigue score after the ERCP | half a year
  fatigue were measured on a 0-10VAS at arrival in the recovery room ,30min later

CONTACTS AND LOCATIONS:
Overall Officials: yanqing li, Study Chair — Qilu Hospital of Shandong University
Locations (2):
- China (2):
  - Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan

REFERENCES:
- [Derived] Liu J, Liu X, Peng LP, Ji R, Liu C, Li YQ. Efficacy and safety of intravenous lidocaine in propofol-based sedation for ERCP procedures: a prospective, randomized, double-blinded, controlled trial. Gastrointest Endosc. 2020 Aug;92(2):293-300. doi: 10.1016/j.gie.2020.02.050. Epub 2020 Mar 7. PMID 32156544